CLINICAL TRIAL: NCT02332252
Title: Electrocautery Versus Scalpel for Surgical Skin Incisions in Cesarean Section. A Randomized Controlled Trial.
Brief Title: Electrocautery Versus Scalpel for Surgical Skin Incisions in Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2014-10
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Wound Infection; Electrocautery; Scalpel
MeSH Terms: conditions — Surgical Wound Infection | interventions — Laser Therapy; Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scalpel (Active Comparator): Skin incision performed with a scalpel during cesarean section.
  Interventions: Device: Scalpel; Procedure: Skin incision
- Electrocautery (Experimental): Skin incision performed with an electrocautery during cesarean section.
  Interventions: Device: Electrocautery; Procedure: Skin incision

INTERVENTIONS:
Device: Scalpel — Skin incision performed with a scalpel during cesarean section.
  Arms: Scalpel
Device: Electrocautery — Skin incision performed with an electrocautery during cesarean section.
  Arms: Electrocautery
Procedure: Skin incision

SUMMARY:
To determine the risk of surgical site infection after surgical skin incision, comparing electrocautery vs. scalpel.

ELIGIBILITY:
Inclusion Criteria:

* Elective Cesarean section, regardless of gestational age.

Exclusion Criteria:

* Skin infection in the cesarean section area.
* Emergency cesarean section.
* Presence of a maternal pathology that increases the risk of infection (immunocompromised state).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | 8 days
  Presence of signs of surgical site infection after cesarean section.

SECONDARY OUTCOMES:
Post operative pain | 8 days
  Post operative pain using a visual scale after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Panama